CLINICAL TRIAL: NCT02963545
Title: Simultaneous Assessments of Serotonin and Kynurenine Pathways Parameters in Patients Shortly (Less Than 4 Hours and a Half) After the Onset of a Cerebral Infarction
Brief Title: TSK (Tryptophan - Serotonin - Kynurenine) Biomarkers Assessment in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Odile VAROQUAUX, Investigator coordinator, Versailles Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P11/25_AVC-TSK
Record Dates: First submitted 2016-09-16; First posted 2016-11-15 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Cerebral Infarction
MeSH Terms: conditions — Cerebral Infarction | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients presenting cerebral infarction (Experimental): no intervention of health product administration,
  Interventions: Other: Usual care patients in neurology department; Biological: blood and urines sampling; Procedure: Psychiatric evaluation
- Historical controls (Other): no intervention of health product administration, patients characteristics, history, matched with patients for age, gender, tobacco consumption and season of inclusion, free of neurologic or psychiatric disease or psychotropic medications or medications known to impact on serotonin
  Interventions: Biological: blood and urines sampling

INTERVENTIONS:
Other: Usual care patients in neurology department — patients characteristics, history, clinical signs chronology and usual medical care by the emergency units, cerebral infarction area
  Arms: Patients presenting cerebral infarction
Biological: blood and urines sampling — Collection samples for biochemical determinations of serotonin pathway and kynurenine pathway parameters determinations
Procedure: Psychiatric evaluation — depression scale, impulsivity scale, hostility scale , tobacco consumption questioning
  Arms: Patients presenting cerebral infarction

SUMMARY:
Single-center, prospective, descriptive and biomedical research with controls, without health product.

Depression is the second risk factor for stroke as tobacco smoking following hypertension. Peripheral abnormalities in serotonin parameters were described in depression and tobacco smoking. The investigators hypothesized dysregulations in pathways of serotonin (5-HT), which has notably complex vasomotor effects and of kynurenine which could have cognitive dysfunction effects.

The aim of this study is to evaluate simultaneously the involvement of serotonin and kynurenine pathways parameters in patients suffering from a cerebral infarction shortly after the onset (less than 4 hours and a half), within a 2 days follow-up (Day 1 and Day 2) and 3 months after the cerebral infarction.

DETAILED DESCRIPTION:
Tryptophan (TRP), an essential aminoacid, is metabolized in the serotonin (5-HT) or in the kynurenine (KYN) pathway. Serotonin is catabolized to 5-HIAA (5-hydroxyindole amino acid) by monoamine oxidase A (MAOA). The TRP to KYN transformation is regulated by indoleamine 2,3-dioxygenase (IDO).

The primary objective was the measurements of serotonin and kynurenine pathways parameters which were performed in blood and urine samples using different HPLC techniques and of serotonin transporters and receptors which were determined in blood platelets. The results in patients were compared to those measured in controls matched for age, gender, tobacco consumption and season of inclusion.

The secondary objective was to evaluate the potential relationships between these 5-HT and Kyn pathways biomarkers concentrations, MAOA and IDO enzymatic activations and clinical outcome and criteria.

ELIGIBILITY:
Study population : patients who had positive MRI diagnosis of cerebral infarction less than 4.30 hours after the clinical onset.

Experimental group :

Inclusion Criteria:

* Age ≥ 18 ans
* Cerebral infarction with a medical care to emergencies less than 4.30 hours after the symptoms onset.
* Written informed consent signed by the patient, or by a trusted person then by the patient himself if permitted by his condition.

Exclusion Criteria:

* Cerebral infarction with a medical care to emergencies more than 4.30 hours after the symptoms onset.
* Patient with subarachnoid haemorrhage, cerebral hematoma.
* Pregnant woman
* Patient under guardianship or trusteeship, or safeguard justice.

Control group :

* Matching criteria for age, gender, tobacco smoking, inclusion season

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Measure of serotonin pathway parameters concentrations in blood and urine samples | Day 1
  platelet serotonin (nM), plasma serotonin (nM), urine serotonin (nM) , plasma 5-HIAA (nM) , urine 5-HIAA (nM) concentrations using three different HPLC systems and methods.
Measure of serotonin pathway parameters in blood samples | Day 1
  Blood platelets assessements of serotonin (5-HT) transporters using [3H]paroxetine ligand ( fmol/mg proteins) and 5-HT2A receptors using [3H]MDL-100,907 ligand ( fmol/mg proteins)
Measure of serotonin pathway parameters in blood and urine samples | Day 2
  platelet serotonin (nM), plasma serotonin (nM), urine serotonin (nM) , plasma 5-HIAA (nM) , urine 5-HIAA (nM) concentrations using three different HPLC systems and methods
Measure of serotonin pathway parameters in blood and urine samples | Month 3
  platelet serotonin (nM), plasma serotonin (nM), urine serotonin (nM) , plasma 5-HIAA (nM) , urine 5-HIAA (nM) concentrations using three different HPLC systems and methods
Measure of kynurenin pathway parameters in blood samples | Day 1
  The first and regulatory enzyme of the kynurenine pathway is the indoleamine-2,3-dioxygenase (IDO). Plasma tryptophan (µM) and plasma kynurenine (µM) concentrations [Trp] and [Kyn] were quantified with HPLC method. [Trp] / [Kyn] ratio (in AU, Arbitrary Units) was used as index for IDO activity .
Measure of kynurenin pathway parameters in blood samples | Day 2
  The first and regulatory enzyme of the kynurenine pathway is the indoleamine-2,3-dioxygenase (IDO). Plasma tryptophan (µM) and plasma kynurenine (µM) concentrations [Trp] and [Kyn] were quantified with HPLC method. [Trp] / [Kyn] ratio (in AU, Arbitrary Units) was used as index for IDO activity .
Measure of kynurenin pathway parameters in blood samples | Month 3
  The first and regulatory enzyme of the kynurenine pathway is the indoleamine-2,3-dioxygenase (IDO). Plasma tryptophan (µM) and plasma kynurenine (µM) concentrations [Trp] and [Kyn] were quantified with HPLC method. [Trp] / [Kyn] ratio (in AU, Arbitrary Units) was used as index for IDO activity .

OTHER OUTCOMES:
Patient characteristics, history, clinical signs chronology | Day 1
  For patients: patient characteristics, history, clinical signs chronology and medical care by pre-hospital then hospital neurology intensive care, MRI diagnosis validation, cerebral infarction area.
  For controls : patient characteristics, history.
Patient characteristics, clinical signs | Day 2
  patients characteristics, clinical signs and medical care by hospital neurology intensive care.
Patient characteristics, clinical signs | Month 3
  Patients characteristics, clinical signs and medical care.
  .
Depression scale | Day 2
  Interview with the patient, or a patient closely related, or a physician. Scale for depression scores (simplified depression scale from Whooley 2006), concerning the 2 weeks before stroke
Impulsivity scale | Day 2
  Interview with the patient, or a patient closely related, or a physician. Scale for impulsivity scores ( Barratt Impulsiveness scale), concerning the 2 weeks before stroke

CONTACTS AND LOCATIONS:
Overall Officials: Odile SPREUX-VAROQUAUX, PhD, Principal Investigator — Pharmacology, Versailles Hospital and Versailles University; Fernando PICO, Neurology Department head, Study Director — Versailles Hospital
Locations (1):
- Centre Hospitalier de Versailles, Le Chesnay, France